CLINICAL TRIAL: NCT04636970
Title: Unobtrusive Technologies for Monitoring of Autonomic Nervous System Function in a Setting of Inpatient Cardiac Rehabilitation and Home Training Program in Elderly Patients With Different Frailty Stages
Brief Title: Unobtrusive Technologies for Monitoring of Autonomic Nervous System Function in Elderly Frail Patients
Acronym: FrailHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Kaunas University of Technology (Other)
Responsible Party: Principal Investigator, Eglė Tamulevičiūtė-Prascienė, Head of a Rehabilitation department, Lithuanian University of Health Sciences hospital Kaunas Clinics, Kulautuva rehabilitation hospital, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUHS002
Record Dates: First submitted 2020-11-09; First posted 2020-11-19 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Frailty; Autonomic Nervous System Imbalance
Keywords: Cardiac rehabilitation; Cardiac surgery; Resistance training; Exercise training; Frailty; Elderly
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients randomised to control group will get usual recommendations regarding physical activity after a discharge from inpatient cardiac rehabilitation.
- Intervention group (Experimental): Patients randomised to intervention group will continue home exercise training that will last 12 weeks and consists of endurance, flexibility, balance and cardiovascular resistance training performed with low to moderate intensity, in 20-60 minutes sessions, five times a week. Study participants will be asked to wear wrist and chest unobtrusive devices during active day time or at least during the training session and two hours before and after. Study participants well receive telephone calls every other week and were asked to answer questions regarding their health and physical activity.
  Interventions: Other: Home training program

INTERVENTIONS:
Other: Home training program — Subjects randomized to the IG will participate at home training program that will last 12 weeks and consists of endurance, flexibility, balance and cardiovascular resistance training performed with low to moderate intensity, in 20-60 minutes sessions, five times a week. Study participants will be asked to wear wrist and chest unobtrusive devices during active day time or at least during the training session and two hours before and after.
  Arms: Intervention group

SUMMARY:
To develop and investigate an unobtrusive technology for long-term monitoring of autonomic nervous system (ANS) function's response to daily physical stressors and exercise training for elderly patients with different frailty stages.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to CR after open heart surgery.
* Age 65 years and older.
* 6-minute walk distance (6-MWD) ≥150 meters.
* Patient's agreement to participate in the study.
* Edomonton Frailty Scale score 5 points and more

Exclusion Criteria:

* Cardiac devices (due to artificially altered heart rate series)
* Diseases in the musculoskeletal system or other organs complicating physical activity and exercise training;
* Exercise-limiting comorbidities (primarily orthopedic and neurological conditions that would exclude individuals from participating in CR according to study protocol), including chronic heart failure New York Heart Association Class IV, hemoglobin less than 9 g/dL, wound healing disturbance, cognitive or linguistic deficits.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Autonomic nervous function by Heart Rate Recovery (HRR) | 3 weeks
  HRR (beats per minute) is a difference of the maximal HR obtained during stress testing and HR during the recovery period: HR30-360 the decay of heart rate from 30 to 360 s after the recovery onset.
Autonomic nervous function by Heart Rate Recovery (HRR) | 12 weeks
  HRR (beats per minute) is a difference of the maximal HR obtained during stress testing and HR during the recovery period: HR30-360 the decay of heart rate from 30 to 360 s after the recovery onset.
Autonomic nervous function by Heart Rate Fragmentation (HRR) | 3 weeks
  HRF measured by RR interval indexes:percentage of inflection points (PIP), inverse of the average length of the acceleration/deceleration segments (IALS), percentage of short segments (PAS), percentage of alternation segments (PSS).
Autonomic nervous function by Heart Rate Fragmentation (HRR) | 12 weeks
  HRF measured by RR interval indexes:percentage of inflection points (PIP), inverse of the average length of the acceleration/deceleration segments (IALS), percentage of short segments (PAS), percentage of alternation segments (PSS).

SECONDARY OUTCOMES:
Cardiopulmonary exercise capacity by maximal oxygen consumption (peakVO2) | 3 weeks
  PeakVO2 measured with spiroergometry by millilitres of oxygen per kilogram of body mass per minute
Cardiopulmonary exercise capacity by maximal oxygen consumption (peakVO2) | 12 weeks
  PeakVO2 measured with spiroergometry by millilitres of oxygen per kilogram of body mass per minute
Cardiopulmonary exercise capacity by maximal load (maxWatt) | 3 weeks
  Maximal load measured with spiroergometry by maximal watts
Cardiopulmonary exercise capacity by maximal load (maxWatt) | 12 weeks
  Maximal load measured with spiroergometry by maximal watts
Functional capacity by six minutes walking test (6MWT) | 3 weeks
  6MWT measured by meters
Functional capacity by six minutes walking test (6MWT) | 12 weeks
  6MWT measured by meters
Physical performance by Timed up and Go test (TUG) | 3 weeks
  TUG measured by seconds
Physical performance by Timed up and Go test (TUG) | 12 weeks
  TUG measured by seconds
Gait evaluation by step time | 3 weeks
  Step time measured with treadmill ergometer by seconds
Gait evaluation by step time | 12 weeks
  Step time measured with treadmill ergometer by seconds
Frailty level by Edmonton frailty scale (EFS) | 3 weeks
  0-17 points, the higher the worse. The EFS assesses 9 domains: cognition, general health status, functional independence, social support, medication use, nutrition, mood, continence, and functional performance.
Frailty level by Edmonton frailty scale (EFS) | 12 weeks
  0-17 points, the higher the worse. The EFS assesses 9 domains: cognition, general health status, functional independence, social support, medication use, nutrition, mood, continence, and functional performance.

CONTACTS AND LOCATIONS:
Overall Officials: Raimondas Kubilius, MD, PhD, Principal Investigator — Lithuanian University of Health Sciences, Department of Rehabilitation
Locations (1):
- LUHS hospital Kaunas Clinics Rehabilitation hospital of Kulautuva, Kaunas, Kulautuva, Lithuania

IPD SHARING:
Plan to Share IPD: No
Individual participant anonymous data may be shared upon appropriate request.